CLINICAL TRIAL: NCT06641778
Title: Fecal Microbiota Transplantation in Patients With Multiple Drug Resistant Klebsiella Pneumoniae Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: luxia Kong (Other)
Responsible Party: Sponsor-Investigator, luxia Kong, physician, Wuhan Central Hospital
Organization: Wuhan Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LXKong
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Klebsiella Pneumoniae Pneumonia
Keywords: Fecal Microbiota Transplantation; Multiple Drug Resistant Klebsiella Pneumoniae Pneumonia
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group of patients received conventional antibiotic therapy and fecal microbiota transplantation.
  Interventions: Other: Fecal Microbiota Transplantation
- control group (No Intervention): Patients in this group were treated with conventional antibiotics.

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Patients in the experimental group received conventional antibiotic therapy plus fecal microbiota transplantation, and the efficacy was compared with that in the control group
  Arms: experimental group

SUMMARY:
Multidrug-resistant Klebsiella pneumoniae (MDR-KP) infections account for 10% of all nosocomial infections, and even with effective antibiotics, the mortality rate is as high as 50%. Intestinal bacteria transplantation can not only treat intestinal diseases, but also inhibit the colonization and proliferation of drug-resistant bacteria. This study explored the therapeutic value of fecal microbiota transplantation in patients with MDR-KP pneumonia.

DETAILED DESCRIPTION:
Intervention study (controlled clinical study) : patients with multidrug-resistant Klebsiella pneumoniae pneumonia were randomly assigned to the experimental group (conventional antibiotic treatment + fecal microbiota transplantation) and the control group (conventional antibiotic treatment); The clinical symptoms, inflammatory indexes, immune indexes, intestinal microecology, respiratory microecology and antibiotic resistance gene changes were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Meet the diagnostic criteria for community-acquired pneumonia or hospital-acquired pneumonia;
* The etiological results of sputum or alveolar lavage fluid suggested MDR-KP infection;
* The patient or his family members voluntarily participated, collected alveolar lavage fluid and stool samples, agreed to perform FMT treatment, and signed the informed consent.

Exclusion Criteria:

* Subjects with persistent bronchial asthma, severe pulmonary dysfunction, or inability to tolerate bronchoscopy;
* Patients with severe damage of intestinal barrier such as sepsis and digestive tract perforation due to various reasons;
* Those currently diagnosed with explosive colitis or toxic megacolon have gastroesophageal reflux disease or peptic ulcer; Subjects taking probiotics within 6 months;
* Enteral nutrition patients who could not tolerate 50% of heat calorie requirements due to severe diarrhea, significant fibrous intestinal stenosis, severe gastrointestinal bleeding, high-flow intestinal fistula and other reasons.
* Patients with obvious bleeding tendency, severe pulmonary hypertension, superior vena cava obstruction, and aortic aneurysm rupture risk;
* Patients with malignant hypertension, recent myocardial infarction (≤6 months), severe arrhythmia, and cardiac insufficiency;
* suffering from malignant tumor diseases, congenital or acquired immune deficiency diseases, other systemic inflammatory response diseases;
* Those who have recently been treated with high-risk immunosuppressive/cytotoxic drugs, such as rituximab, doxorubicin, or steroid hormones (20mg/d ponisone or higher) for more than 4 weeks;
* Severe immunosuppression: adult neutrophils <1 500/mm3, child neutrophils <1 000/mm3;
* Pregnancy or lactation;
* There is a mental disability or active mental illness that prevents informed consent;
* Conditions deemed unsuitable for study inclusion by other clinicians.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of days MDR-KP turns negative | one month
  The number of days that multidrug-resistant Klebsiella pneumoniae turned negative after treatment
Length of hospital stay | one month
  Total length of stay from admission to discharge or death
mortality rate | one month
  The ratio of death cases to the total number of patients

SECONDARY OUTCOMES:
The Incidence of fever | one month
  The incidence of fever in patients was included
The incidence of cough | one month
  The incidence of cough in patients was included
The incidence of phlegm | one month
  The incidence of phlegm in patients was included
The incidence of chest pain assessed by VAS | one month
  The incidence of chest pain in patients was included

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Geng, Study Director — Wuhan Central Hospital
Locations (1):
- The central Hospital of Wuhan, Wuhan, Hubei, China